CLINICAL TRIAL: NCT01576861
Title: Long-Term Efficacy and Safety of Growth Hormone Replacement Therapy in Chronic Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Antonio Cittadini, Associate Professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Long-Term GH in CHF
Record Dates: First submitted 2012-03-19; First posted 2012-04-13 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Growth Hormone Deficiency; Chronic Heart Failure
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Growth Hormone

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- GH replacement (Experimental): Patients will receive 48 months of substitutive somatotropin (growth hormone) therapy at a dose of 0,012 mg/kg every second day, added to their background optimized CHF therapy
  Interventions: Drug: Somatotropin
- Control CHF patients under optimized CHF therapy (No Intervention)

INTERVENTIONS:
Drug: Somatotropin — Subcutaneous Somatotropin (recombinant Human Growth Hormone) 0,012 mg/kg every second day
  Arms: GH replacement

SUMMARY:
After the encouraging results of 6 months of Growth Hormone Replacement Therapy in Patients With Chronic Heart Failure and Coexisting Growth Hormone Deficiency (NCT00591760) the investigators wanted to collect data about the long-term efficacy and safety of this kind of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Heart Failure New York Heart Association functional class II to IV, secondary to ischemic or idiopathic cardiomyopathy
* Age range 18-80 years
* Stable medication for at least one month including beta-blockers that had to be started at least 5 months before entering the study
* Left Ventricular ejection fraction 40% or less
* Growth Hormone Deficiency (defined as a peak GH response to intravenous stimulation with GHRH + Arginine < 9 ng/ml)
* Written Informed consent

Exclusion Criteria:

* Acute proliferative or severe non-proliferative diabetic retinopathy
* Active malignancy
* Evidence of progression or recurrence of an underlying intracranial tumor
* Unstable Angina or recent myocardial infarction
* Serum Creatinine levels > 2.5 mg/dl
* Severe liver disease (Child-Pugh B-C)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-01; Primary Completion 2011-03 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Peak Oxygen Consumption | after 48 months
Side effects | Any side effects recorded after 6,24 and 48 months

SECONDARY OUTCOMES:
Left Ventricular Ejection Fraction | after 48 months
Left Ventricular End-Systolic Volume | after 48 months
Left Ventricular End-Diastolic Volume | after 48 months
Quality of Life | after 48 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Cardiovascular and Immunological Sciences, Napoli, Campania, Italy